CLINICAL TRIAL: NCT03672864
Title: Parent Therapist Partnership to Provide Early, Intensive Exercise to Enhance Walking Outcomes in Children With Perinatal Stroke
Brief Title: Parent Therapist Partnership to Provide Early, Intensive Exercise in Perinatal Stroke
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Brain Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00078553
Record Dates: First submitted 2018-09-13; First posted 2018-09-17 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Perinatal Stroke
Keywords: Walking; Intensive exercise; Rehabilitation; Cerebral Palsy; Early intervention
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: Randomized, controlled trial
Who Masked: Outcomes Assessor
Masking Description: Assessing therapists are masked to the child's group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate Group (Experimental): The intervention is intensive exercise, delivered over 12 weeks beginning on admission to the study. The group will then be followed for 9 months post intervention.
  Interventions: Behavioral: Intensive exercise
- Delay Group (No Intervention): The group will be followed for 6 months with no intervention. After 6 months the group will be given the opportunity to receive the same intensive exercise intervention as the Immediate group. The group will be followed for 3 months following the intervention.

INTERVENTIONS:
Behavioral: Intensive exercise — Intensive, child-initiated movement of the lower extremity: 1 hour/day, 4 days/week, 2 sessions delivered by a physical therapist, 2 delivered by a parent. All activities are play based, and exercise intensity is enhanced by small weights placed on the dorsum of the foot and the ankle of the affected limb. Intervention is delivered over 12 weeks for a target of 48 hours of training.
  Arms: Immediate Group

SUMMARY:
A prospective, single blind, parallel group, randomized control trial to determine if early, intensive lower extremity activity delivered by a physical therapist and a parent in partnership improves gross motor function more than usual care.

DETAILED DESCRIPTION:
A mixed-methods randomized controlled trial at 3 healthcare centres: Edmonton, Calgary and Ottawa. The period of participation for each child is 12 months. The Immediate Group will have 3 months of intervention and 9 months follow-up. The Delay Group will be followed for 6 months (waitlist-control period), then given the opportunity to receive the same intervention and followed for 3 months after the intervention.

The intervention will be delivered by clinicians in the rehabilitation centres in partnership with the child's parents. Therapists will provide training 2 days a week and will coach the parents to provide the training at home for 2 days a week.

The intervention is ELEVATE (Engaging the Lower Extremity Via Active Therapy Early) and consists of child-initiated, intensive leg activities for one hour a day, four days a week for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* children ages 8 months to 3 years
* medical history and physical exam consistent with perinatal stroke
* hemiparesis in the upper and/or lower extremity
* parental agreement to adhere to the training and testing schedule

Exclusion Criteria:

* bilateral motor impairment
* epileptic seizures that could interfere with training
* cognitive, behavioural or developmental impairments that preclude participation in the protocol
* botulinum toxin A injections or surgery in the lower extremities within the previous six months
* concurrent casting during the intervention phase (including constraint-induced movement therapy with casting)
* diagnosis associated with neurological/developmental regression
* parent unable to communicate (verbal and written) in English or French

Ages: 8 Months to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 18 (Actual)
Dates: Start 2019-02-15 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Gross Motor Function Measure (GMFM-66) - change from baseline | 3 months, 6 months, 9 months, 12 months
  A 66 item criterion referenced observational measure of gross motor skills designed for children with cerebral palsy.

SECONDARY OUTCOMES:
The Pediatric Quality of Life Measure module for cerebral palsy (PedsQL CP) - change from baseline | 3 months, 6 months, 9 months, 12 months
  A questionnaire completed by parents including 5 scales: 1) daily activities, 2) movement and balance, 3) pain and hurt, 4) fatigue, and 5) eating activities.
Ankle joint angle at onset of stretch reflex - change from baseline | 3 months, 6 months, 9 months, 12 months
  Ankle joint angle caused by the stretch reflex will be measured with the Portable Spasticity Assessment Device (PSAD). A hand-held segment of the device is applied to the foot segment to measure the motion of the limb. Disposable, surface electromyographic electrodes are applied to the skin of the limb to measure the muscle activity.
Ankle joint angle at full dorsiflexion - change from baseline | 3 months, 6 months, 9 months, 12 months
  Ankle joint angle at the extreme of dorsiflexion will be measured with the Portable Spasticity Assessment Device (PSAD). A hand-held segment of the device is applied to the foot segment to measure the motion of the limb. Disposable, surface electromyographic electrodes are applied to the skin of the limb to ensure the muscle is relaxed during the measurement.
Resource use questionnaire | Baseline
  All health, community, and social service use will be collected at baseline and every six months throughout the one year study period using the Resource Use Questionnaire, a tool validated for use in participants with neurodevelopmental disabilities. Costs related to lower extremity therapy as well as resources used for treatment and management of the child's cerebral palsy will be included over the study period.
Resource use questionnaire | 6 months
  All health, community, and social service use will be collected at baseline and every six months throughout the one year study period using the Resource Use Questionnaire, a tool validated for use in participants with neurodevelopmental disabilities. Costs related to lower extremity therapy as well as resources used for treatment and management of the child's cerebral palsy will be included over the study period.
Resource use questionnaire | 12 months
  All health, community, and social service use will be collected at baseline and every six months throughout the one year study period using the Resource Use Questionnaire, a tool validated for use in participants with neurodevelopmental disabilities. Costs related to lower extremity therapy as well as resources used for treatment and management of the child's cerebral palsy will be included over the study period.
Young Children's Participation and Environment Measure (YC-PEM) - change from baseline | 3 months, 6 months, 9 months, 12 months
  A questionnaire completed by parents to assess participation in three settings: home, daycare/preschool, and the community.

OTHER OUTCOMES:
Qualitative study using Interpretative Description methodology | Immediately before and after the intervention
  A concurrent qualitative study will be conducted to gain insight into the perspective of parents participating in the administration of the ELEVATE intervention and their experiences as a partner in the early, intensive rehabilitation. Semi-structured, individual interviews will be conducted by a researcher with a subset of parents.

CONTACTS AND LOCATIONS:
Overall Officials: Jaynie Yang, Principal Investigator — University of Alberta
Locations (3):
- Canada (3):
  - Alberta Children's Hospital, Calgary, Alberta
  - University of Alberta, Edmonton, Alberta
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hurd CL, Barnes M, Diot CM, Condliffe EG, Alazem H, Pritchard L, Zwicker JD, McCormick A, Watt MJ, Andersen J, Kirton A, Yang JF. Parent-therapist partnership to ELEVATE gross motor function in children with perinatal stroke: protocol for a mixed methods randomized controlled trial. BMC Pediatr. 2022 Aug 10;22(1):480. doi: 10.1186/s12887-022-03525-6. PMID 35948896